CLINICAL TRIAL: NCT05549726
Title: A Multisectoral Strategy to Address Persistent Drivers of the HIV Epidemic in East Africa: SEARCH CAB LA Dynamic Choice HIV Prevention Study Extension
Brief Title: SEARCH CAB LA Dynamic Choice HIV Prevention Study Extension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); Makerere University (Other); Kenya Medical Research Institute (Other); University of California, Berkeley (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); ViiV Healthcare (Industry); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEARCH CAB LA Extension; U01AI150510 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: Cabotegravir Injectable Suspension; PrEP; HIV Treatment and Prevention; Community Health
MeSH Terms: interventions — cabotegravir; Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants initially randomized to the Dynamic Choice Prevention delivery model will be given the option to use CAB-LA as part of the dynamic choice prevention delivery package. Participants initially randomized to standard of care will continue to receive standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dynamic choice prevention (including CAB LA) (Experimental): The Dynamic Choice Delivery Model includes integrated PrEP and PEP services at outpatient clinics, antenatal clinics, and via VHT workers in community households. CAB-LA will be integrated into the dynamic choice delivery model as an additional biomedical prevention option in a patient-centered delivery model based on the precede framework.
  Interventions: Drug: Cabotegravir Injectable Suspension; Other: Dynamic Choice Delivery Model
- Standard of Care (Active Comparator): The standard of care for PEP or PrEP differs according to each country's guidelines.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Cabotegravir Injectable Suspension — CAB-LA will be one of the options for the Dynamic Choice Delivery intervention arm. CAB-LA will be a choice for at-risk adults and adolescents weighing at least 35 kg for pre-exposure prophylaxis (PrEP) to reduce the risk of sexually acquired HIV-1 infection. Single-dose vial containing 600 mg/3 mL (200 mg/mL) of cabotegravir is a white to light pink, free-flowing, extended-release injectable suspension. CAB-LA administration will occur at health facilities.
  Arms: Dynamic choice prevention (including CAB LA)
Other: Dynamic Choice Delivery Model — The Dynamic Choice Delivery Model includes integrated PrEP (including CAB-LA) and PEP services at outpatient clinics, antenatal clinics, and via VHT workers in community households. The procedures for each trial include PrEP/PEP counseling and services, choice of service location, HIV testing options, option for longer PrEP refills, provision of a clinical officer's or nurse's mobile telephone number for immediate PEP starts any day of the week, assessment of PrEP/PEP barriers and personalized actions, psychologic supports for traumatic experiences, and offer of concurrent, additional health or prevention related services.
  Arms: Dynamic choice prevention (including CAB LA)
Other: Standard of Care — The standard of care differs according to country but does not routinely offer PEP or PrEP to clients seeking services, does not offer choice of service location, HIV testing option or access to medical provider mobile phone number.
  Arms: Standard of Care

SUMMARY:
The overall purpose of this SEARCH CAB-LA (Cabotegravir Injectable Suspension) randomized extension study is to determine if adding the option of CAB-LA as a prevention choice using a person-centered dynamic choice HIV (human immunodeficiency virus) prevention model, with option to switch products over time, compared to the standard of care: 1) increases prevention coverage; 2) reduces HIV incident infection; and 3) increases prevention coverage during periods of self-assessed risk of HIV infection, in three settings in rural Uganda and Kenya.

In addition, this study will describe implementation of a person-centered model for dynamic choice HIV prevention including CAB-LA, using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) evaluation framework among persons randomized to the intervention arm.

DETAILED DESCRIPTION:
The SEARCH CAB-LA (Cabotegravir Injectable Suspension) dynamic choice HIV prevention study is a randomized extension study of a person-centered Dynamic Choice HIV Prevention model for delivering existing evidence-based biomedical prevention interventions vs. standard of care (SOC). The study is conducted in 3 settings in rural Western Uganda and Kenya: antenatal (ANC) clinics, the outpatient department (primary care clinics), and in community settings. Participants previously randomized to Dynamic Choice HIV Prevention or SOC are re-consented and remain in their initial randomized arm. During the extension, the Dynamic Choice HIV Prevention intervention offers participants choices of biomedical prevention product (oral Pre-Exposure Prophylaxis (PrEP), oral post-exposure prophylaxis (PEP), or Cabotegravir Injectable Suspension (CAB-LA) on an ongoing basis with the option to switch products over time based on participant preference and perceived risk. The primary endpoint is proportion of time that is covered by a biomedical prevention product over 48 weeks; secondary endpoints are: i) incident HIV infection over 48 weeks; and, ii) proportion of time during which a participant reports risk of HIV infection that is covered by a biomedical prevention product over 48 weeks. Participants in the intervention arm only are reconsented at 48 weeks for implementation evaluation up to 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the Extension include:

1. Enrollment in a SEARCH Sapphire Dynamic prevention study (NCT04810650)
2. HIV negative at start of extension
3. Residing in study region

Additional inclusion criteria to access CAB-LA as a prevention option

1. Not pregnant or breastfeeding at time of initial CAB-LA injection
2. Participant weighs at least 35kg

Exclusion Criteria:

Exclusion criteria to access CAB-LA as a prevention option:

1. Participant has Hepatitis B or chronic Hepatitis C Diagnosis
2. Participant has ALT >=5x ULN
3. Participant has clinical history of liver cirrhosis or current clinical evidence of cirrhosis
4. Previous hypersensitivity reaction to cabotegravir
5. Receiving the following co-administered drugs for which significant decreases in cabotegravir plasma concentrations may occur due to uridine diphosphate glucuronosyltransferase:

   i. Anticonvulsants: Carbamazepine, oxcarbazepine, phenobarbital, phenytoin ii. Antimycobacterials: Rifampin, rifapentine
6. Participants with a current or anticipated need for chronic systemic anticoagulation or a history of known or suspected bleeding disorder, including a history of prolonged bleeding, except for the use of anticoagulation for deep vein thrombosis (DVT) prophylaxis (e.g., postoperative DVT prophylaxis) or the use of low dose acetylsalicylic acid (≤325 mg).

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Principal Investigator — University of California, San Francisco; Moses Kamya, MBChB, PhD, Principal Investigator — Makerere University; Maya Petersen, MD, PhD, Principal Investigator — University of California, Berkeley
Locations (2):
- GPRT / SEARCH Office, Kisumu, Kenya
- IDRC Southwest Uganda, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamya MR, Balzer LB, Ayieko J, Kabami J, Kakande E, Chamie G, Sutter N, Sunday H, Litunya J, Schwab J, Schrom J, Bacon M, Koss CA, Rinehart AR, Petersen M, Havlir DV; SEARCH Consortium. Dynamic choice HIV prevention with cabotegravir long-acting injectable in rural Uganda and Kenya: a randomised trial extension. Lancet HIV. 2024 Nov;11(11):e736-e745. doi: 10.1016/S2352-3018(24)00235-2. Epub 2024 Oct 9. PMID 39395424

RESULTS

PARTICIPANT FLOW:
Groups:
- Dynamic Choice Prevention (Including CAB LA): The Dynamic Choice Delivery Model includes integrated PrEP and PEP services at outpatient clinics, antenatal clinics, and via VHT workers in community households. CAB-LA will be integrated into the dynamic choice delivery model as an additional biomedical prevention option in a patient-centered delivery model based on the precede framework.
  Cabotegravir Injectable Suspension: CAB-LA will be one of the options for the Dynamic Choice Delivery intervention arm. CAB-LA will be a choice for at-risk adults and adolescents weighing at least 35 kg for pre-exposure prophylaxis (PrEP) to reduce the risk of sexually acquired HIV-1 infection. Single-dose vial containing 600 mg/3 mL (200 mg/mL) of cabotegravir is a white to light pink, free-flowing, extended-release injectable suspension. CAB-LA administration will occur at health facilities.
  Dynamic Choice Delivery Model: includes integrated PrEP (including CAB-LA) and PEP services at outpatient clinics, antenatal clinics, and via VHT workers in community households. The procedures for each trial include PrEP/PEP counseling and services, choice of service location, HIV testing options, option for longer PrEP refills, provision of a clinical officer's or nurse's mobile telephone number for immediate PEP starts any day of the week, assessment of PrEP/PEP barriers and personalized actions, psychologic supports for traumatic experiences, and offer of concurrent, additional health or prevention related services.
Period: Overall Study
Arm/Group | Dynamic Choice Prevention (Including CAB LA) | Standard of Care
Started | 487 | 497
Completed | 485 | 492
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dynamic Choice Prevention (Including CAB LA) | Standard of Care | Total
Number analyzed (Participants) | 487 | 497 | 984
Age, Customized [Count of Participants; unit: Participants]
  Age: 15-24 | 139 | 159 | 298
  Age: >=25 | 348 | 338 | 686
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 358 | 358 | 716
  Male | 129 | 139 | 268
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 487 | 497 | 984
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 242 | 239 | 481
  Kenya | 245 | 258 | 503

OUTCOME MEASURES:

1. Primary Outcome: Biomedical Prevention Covered Time
Description: Number of days participant taking biomedical prevention divided by number of days participant biomedical prevention use measured.
  Biomedical prevention includes PrEP tenofovir disoproxil fumarate/lamivudine (TDF/3TC) or cabotegravir long-acting injectable (CAB-LA) and PEP
Time Frame: 48 weeks
Population: Study Participants at Week 48 with data on biomedical HIV prevention coverage during follow-up of the extension
Measure: Mean (95% Confidence Interval); unit: % of days
Arm/Group | Dynamic Choice Prevention (Including CAB LA) | Standard of Care
Number analyzed (Participants) | 485 | 492
% of days | 69.7 [64.9 to 74.5] | 13.3 [10.2 to 16.3]

2. Secondary Outcome: HIV Incident Infection
Description: HIV incidence rate: number of HIV incident infections divided by number at risk (HIV incidence per 100 person-years)
Time Frame: 48 weeks
Measure: Number; unit: infections per 100 person-years
Groups:
- Dynamic Choice Prevention (Including CAB LA): The Dynamic Choice Delivery Model includes integrated PrEP and PEP services at outpatient clinics, antenatal clinics, and via VHT workers in community households. CAB-LA will be integrated into the dynamic choice delivery model as an additional biomedical prevention option in a patient-centered delivery model based on the precede framework.
  CAB-LA will be one of the options for the Dynamic Choice Delivery intervention arm. CAB-LA will be a choice for at-risk adults and adolescents weighing at least 35 kg for pre-exposure prophylaxis (PrEP) to reduce the risk of sexually acquired HIV-1 infection. Single-dose vial containing 600 mg/3 mL (200 mg/mL) of cabotegravir is a white to light pink, free-flowing, extended-release injectable suspension. CAB-LA administration will occur at health facilities.
  Dynamic Choice Delivery Model: The Dynamic Choice Delivery Model includes integrated PrEP (including CAB-LA) and PEP services at outpatient clinics, antenatal clinics, and via VHT workers in community households. The procedures for each trial include PrEP/PEP counseling and services, choice of service location, HIV testing options, option for longer PrEP refills, provision of a clinical officer's or nurse's mobile telephone number for immediate PEP starts any day of the week, assessment of PrEP/PEP barriers and personalized actions, psychologic supports for traumatic experiences, and offer of concurrent, additional health or prevention related services.
Arm/Group | Dynamic Choice Prevention (Including CAB LA) | Standard of Care
Number analyzed (Participants) | 485 | 486
infections per 100 person-years | 0 | 1.8

3. Secondary Outcome: HIV Incident Infection
Description: HIV incidence rate: number of HIV incident infections divided by person time follow-up
Time Frame: 96 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Biomedical Prevention During Periods of Self Assessed HIV Risk
Description: Number of months participant taking biomedical prevention and at self-assessed risk of HIV infection divided by number of months measured and at risk self-assessed risk of HIV infection
Time Frame: 96 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over 48 weeks.
Description: Adverse Events were captured and classified using the NIAID Adverse Event Grading of Severity scale in the intervention arm. All deaths, life threatening events, hospitalizations, significant disability due to AE, and congenital anomaly/birth defects were classified as SAE regardless of relationship. Grade 3 and 4 and non-serious adverse drug reaction leading to withdrawal were captured for participants on CAB-LA.
Arm/Group | Dynamic Choice Prevention (Including CAB LA) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/487 | 2/497
Serious Adverse Events (participants affected / at risk) | 4/487 | 2/497
Other Adverse Events (participants affected / at risk) | 0/487 | 0/497
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dynamic Choice Prevention (Including CAB LA) (N=487) | Standard of Care (N=497)
Ocular injury (Eye disorders) | 1 (1) | 0 (0)
Hospitalization due to physical altercation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Premature birth and deaths of twins (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Miscarriage following blunt abdominal trauma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Death due to motorcycle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Death due to unknown causes (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Participants maintained their original randomization group; so balance at extension start wasn't guaranteed. Sensitivity analyses adjusted for baseline differences, but unmeasured differences may remain. Self-reported pill ingestion (PrEP/PEP) may have recall bias; CABLA injections were logged. HIV incidence differences validate intervention impact.We relied on self-reported risk without specific classifications and evaluated a combination intervention,complicating effect attribution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT05549726/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT05549726/SAP_001.pdf
  • Informed Consent Form (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT05549726/ICF_002.pdf